CLINICAL TRIAL: NCT05335187
Title: Hybrid Micro-macro Electrodes to Record the Activity of Single Neurons During Seizures in Patients Who Suffer from Epilepsy
Brief Title: Hybrid Micro-macro Electrodes in Patients with Epilepsy
Acronym: MicroEPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Mégevand (Other)
Collaborators: Swiss National Science Foundation (Other); Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Sponsor-Investigator, Pierre Mégevand, Assistant Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-D0033; 194507 (Other Grant/Funding Number: Swiss National Science Foundation); 10001031 (Other: Swissmedic)
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy
Keywords: drug-resistant epilepsy; epilepsy monitoring unit; intracranial EEG; microelectrodes; neuronal recordings; epilepsy surgery
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- micro-macro electrode (Experimental): In this single-arm, open-label study, all patients receive one or a handful of micro-macro electrode (MME) in place of conventional intracranial EEG electrodes.
  Interventions: Device: micro-macro electrode implantation

INTERVENTIONS:
Device: micro-macro electrode implantation — One or a handful of micro-macro electrodes are implanted for 2-4 weeks in patients undergoing epilepsy monitoring with intracranial EEG electrodes.

SUMMARY:
The aim of the MicroEPI study is to know whether it is possible to use safely a medical device (a micro-electrode) that allows recording the activity of neurons in the human brain. Patients who suffer from drug-resistant epilepsy and who are candidates to epilepsy surgery to alleviate their condition sometimes require the implantation of intracranial EEG electrodes for a few weeks, in order to determine as best as possible which region of the brain to operate on. In the MicroEPI study, some of these electrodes will also comprise micro-electrodes, allowing us to record the activity of the patients' neurons during their epileptic seizures.

DETAILED DESCRIPTION:
Epilepsy is a common disease of the brain that can be severe or even cause death. What we call epilepsy is a tendency to suffer from epileptic seizures, which themselves consist in symptoms (e.g. loss of consciousness, involuntary movements, abnormal sensations like hallucinations) caused by abnormally intense or synchronized activity of the brain's neurons. However, we still understand very poorly what exactly goes on at the level of neurons in the human brain during an epileptic seizure. This knowledge gap is due to the fact that the brain's neurons are very small structures and are very well protected by the skull, and are therefore hard to study in human beings. Gaining a better understanding of how neuronal activity goes awry during epileptic seizures could lead to better ways to treat this disease.

In the MicroEPI study, a medical device called micro-macro electrode (MME), manufactured by the company Dixi Medical (France), will be implanted in the brain of patients who must anyway receive intracranial EEG electrodes. These MME electrodes will replace one or a handful of conventional intracranial EEG electrodes. The implantation surgery will be performed in the operating room, under general anesthesia, by an experienced neurosurgeon. The electrodes will remain implanted for 2 to 4 weeks, with the exact duration depending on the time required for the clinical team caring for the patient to collect enough information on the patient's epilepsy. During the entire duration of the electrodes' implantation, the patient will remain hospitalized, and the electrical signals from their brain will be recorded continuously. At the end of this period, the electrodes will be explanted in the operating room. The safety of the MME electrodes, expressed in terms of the number of adverse events attributable to the MME, will be compared to current data on the safety of conventional intracranial EEG electrodes. The performance of the MME electrodes, in terms of the number of recorded neurons, will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or older suffering from drug-resistant focal epilepsy.
* Candidate for epilepsy surgery.
* Requires evaluation with intracranial stereo-EEG electrodes.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Any acute infection (e.g. fever, throat infection).
* Skin or scalp infection over the implantation site.
* Thin or fragile skull bones, which would prevent stereo-EEG electrodes from being anchored safely.
* Increased risk of infections, either from a medical condition or from immunosuppressant medication.
* Increased risk of bleeding, either from a medical condition or from antiplatelet or anticoagulant medication.
* Severe concomitant medical disease (including, but not limited to, cardiovascular, respiratory, renal or hepatic disease).
* Severe concomitant psychiatric disease or major psychological distress.
* Women who are pregnant or breastfeeding during the study.
* Patients who have an implanted stimulation device (e.g. pacemaker, defibrillator, neurostimulator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events (safety outcome) | approximately 30 days
  Number of adverse and severe adverse events possibly, probably or definitely related to the study device

SECONDARY OUTCOMES:
Device malfunctions (performance outcome 1) | approximately 30 days
  Number of device malfunctions preventing the acquisition of microscopic electrophysiological signals
Number of neurons recorded (performance outcome 2) | approximately 30 days
  Number of individual neurons recorded per micro-electrode

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern, Canton of Bern
  - Hôpitaux Universitaires de Genève, Geneva, CH

IPD SHARING:
Plan to Share IPD: Yes
The neurophysiological data will be made available to the research community on an open scientific repository at the study's end.